CLINICAL TRIAL: NCT00945685
Title: Evaluation of Safety and Efficacy of Using Imagine™ Computerized Radiofrequency System for Skin Tightening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endymion Medical Ltd (Industry)
Responsible Party: Dr. Hanna Levy, Endymion Medical Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN-IOP - 01
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Skin Aging; Skin Wrinkling
Keywords: Skin Aging; Skin Wrinkling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endymion study group (Experimental)
  Interventions: Device: Endymion Imagine™ System for Skin Tightening

INTERVENTIONS:
Device: Endymion Imagine™ System for Skin Tightening — Based on patient skin type and area of treatment the physician will choose the following parameters (some parameters are fixed):
  * Pulse energy (J);
  * RF frequency (1MHz);
  * Pulse duration (30 sec);
  * Treatment hand piece (skin tightening);

SUMMARY:
Skin aging is a multifactorial process involving the 3 layers of the skin: Epidermis, dermis and hypodermis. Skin aging process involves among others: skin roughness (epidermis), skin dyschromia (epidermis, dermis), wrinkles and elastosis - skin texture changes due to collagen modification, skin laxity and cellulite (dermis and hypodermis).

EndyMion has developed the Imagine™ system - Computerized Radiofrequency System for Skin Tightening. By using a multielectrodes treatment tip an exact computerized thermal pattern can be produced allowing to selectively heating one or more of the target tissues (epidermis, dermis and hypodermis). In the skin tightening module the dermis and hypodermis would be targeted, creating enough thermal effect to induce collagen remodeling with no ablative thermal damage in the epidermis or dermis. This post marketing study is intended for evaluation of safety and efficacy of the Imagine™ system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females age 30 and up
* Subjects with Fitzpatrick 4 to 9 degrees of elastosis
* Subject able to comprehend and give informed consent for participation in this study
* Subject must commit to all treatments and follow-up visits
* Subject must sign the Informed Consent Form

Exclusion Criteria:

* Subjects with implanted pacemakers, arrhythmias or any other severe known heart disorder
* Subjects with any implantable metal device in the treatment area
* Subjects on any medication that would affect the characteristic of the skin (medical or hormonal), such as "Accutane", within the past 6 months
* Subjects that have had any other invasive or non invasive method of skin therapy or hair removal performed in the past 6 months (in the treated area)
* Subjects who are scheduled or planned for any other invasive or non invasive method of skin therapy or hair removal in the treatment area at the period of the study
* Subjects who have any form of suspicious lesion on the treatment area
* Subjects with history of keloid formations or hypertrophic scarring
* Pregnant or lactating Subjects
* Subjects with Epilepsy or severe migraines
* Subjects with permanent makeup/ tattoo/ body piercing (in the treated area)
* Subjects with any Infection / abscess / pains in treatment target area
* Eczema or dermatitis
* Subjects who suffer from autoimmune disorders or diabetes
* Subjects using blood thinning medications
* Subjects with clotting disorders
* Subjects on drugs or psychologically determined unsuitable for the study
* Subject is suffering extreme general weakness
* Subject objects to the study protocol
* Concurrent participation in any other clinical study
* Physician objection

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The safety of using the Imagine™ System for skin tightening will be established by physician's assessment/observation of adverse events (signs of pain, skin texture alterations or burn). | 3 months

SECONDARY OUTCOMES:
Efficacy endpoint of using the Imagine™ System for skin tightening will be established by level of skin tightness improvement. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Varda Godfried, Dr., Study Director — Endymion Medical Ltd
Locations (1):
- Elman Clinique, Rishon LeZiyyon, Israel